CLINICAL TRIAL: NCT01228526
Title: A Multicenter, Prospective, Observational Study With PriMatrix for the Treatment of Neuropathic Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Mayo Clinic (Other); Samuel Merritt University (Other); New York College of Podiatric Medicine (Other); Temple University (Other); Circleville Foot & Ankle LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: TEI-003
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Foot Ulcers, Diabetic
MeSH Terms: conditions — Foot Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: PriMatrix

SUMMARY:
To evaluate the effectiveness of PriMatrix in the treatment of DFUs in subjects without significantly compromised arterial circulation.

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II diabetes with investigator-confirmed reasonable metabolic control
* Peripheral neuropathy
* A full thickness diabetic plantar foot ulcer of at least 1 cm2 but not exceeding 10 cm2 in area
* An ulcer which has been in existence for a minimum of 30 days, prior to the day of screening

Exclusion Criteria:

* Suspected or confirmed signs/symptoms of wound infection
* Wounds with exposed bone or tendon
* Hypersensitivity to bovine collagen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diabetic foot ulcer and meet the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percent of study ulcers healed | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kavros, DPM, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - California School of Podiatric Medicine at Samuel Merritt University, Oakland, California
  - Mayo Clinic, Rochester, Minnesota
  - New York College of Podiatric Medicine, New York, New York
  - Circleville Foot & Ankle, Circleville, Ohio
  - Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania